CLINICAL TRIAL: NCT02640781
Title: Comparison of Efficacy Between a Newly Designed Covered Stent and Uncovered Stent for Malignant Colorectal Obstruction: a Prospective, Multicenter Study
Brief Title: Comparison of Efficacy Between a Newly Designed Covered Stent and Uncovered Stent for Malignant Colorectal Obstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-2015-0046
Record Dates: First submitted 2015-12-10; First posted 2015-12-29 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- covered stent (Experimental): newly designed covered stent group
  Interventions: Procedure: self-expandable metal stent insertion(covered stent)
- uncovered stent (Active Comparator): currently used uncovered stent group
  Interventions: Procedure: self-expandable metal stent insertion(uncovered stent)

INTERVENTIONS:
Procedure: self-expandable metal stent insertion(covered stent) — Stent insertion was performed by experienced endoscopists under fluoroscopy and by using through-the-scope methods. After the obstructing tumor was identified by endoscopy, a guidewire was introduced through the stricture under endoscopic and fluoroscopic controls. Then, the self-expandable colorectal covered stent delivery catheter was advanced through the working channel of the endoscope over the guidewire until the stent was positioned across the stricture. Upon releasing the stent delivery catheter, stent deployment was initiated proximally and progressed distally. Simple abdominal radiography was performed during and after the procedures to confirm proper stent placement and expansion.
  Arms: covered stent
Procedure: self-expandable metal stent insertion(uncovered stent) — Stent insertion was performed by experienced endoscopists under fluoroscopy and by using through-the-scope methods. After the obstructing tumor was identified by endoscopy, a guidewire was introduced through the stricture under endoscopic and fluoroscopic controls. Then, the self-expandable colorectal stent delivery uncovered catheter was advanced through the working channel of the endoscope over the guidewire until the stent was positioned across the stricture. Upon releasing the stent delivery catheter, stent deployment was initiated proximally and progressed distally. Simple abdominal radiography was performed during and after the procedures to confirm proper stent placement and expansion.
  Arms: uncovered stent

SUMMARY:
Acute colorectal obstruction has been reported to occur in 7 - 29% of all colorectal malignancies, but emergent surgical decompression is associated with high morbidity and mortality rates. Recently, self-expandable metal stents(SEMS) have been suggested as an alternative to surgery and effectively decompress the colonic obstruction and allow for bowel preparation and elective surgery. Theoretically, SEMSs are classified into uncovered stents and covered stents. Covered stents have the advantage of less frequent stent occlusion by tumor in-growth and the disadvantage of a high risk of stent migration, whereas uncovered stents are associated with less stent migration, although they appear to be more prone to tumor ingrowth. To overcome the drawbacks of conventional stents, a double-layered combination covered stent was developed. In the present study, the investigators evaluated the efficacy and safety of the newly designed covered stent by comparing it with the uncovered stent in patients with malignant colorectal obstruction.

ELIGIBILITY:
Inclusion Criteria:

* 20~85-year-old patients with malignant colorectal obstruction either by primary CRC or extracolonic malignancy
* Patients with clinical obstructive symptoms confirmed by CT or colonoscopy

Exclusion Criteria:

* Patients with evidence of bowel perforation or peritonitis
* Cause of obstruction other than malignancy (bowel adhesion or benign stricture)
* Multiple stricture
* Lower rectal cancer obstruction (AV <5cm)

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-12; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Duration of stent patency between stent insertion and recurrence of obstructive symptoms | 2 years after the procedure
  Time between stent insertion and recurrence of obstructive symptoms caused by tumor ingrowth, tumor overgrowth, or stent migration after stent placement

SECONDARY OUTCOMES:
Number of patients with technical success | 2 years after the procedure
  Technical success: Adequate deployment across the entire length of the malignant strictures and proper stent expansion
Number of patients with clinical success | 2 years after the procedure
  Clinical success: Relief from obstructive symptoms as a result of sufficient improvement in stool passage without additional need for endoscopic or surgical re-intervention within 48 hours
Number of patients with complications | 2 years after the procedure
  Complications: stent obstruction, migration, perforation, bleeding, tenesmus, anal pain

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park SJ, Park Y, Lee HJ, Park JJ, Cheon JH, Kim WH, Kim TI. Newly designed flared-end covered versus uncovered self-expandable metallic stents for palliation of malignant colorectal obstruction: a randomized, prospective study. Intest Res. 2025 Apr;23(2):202-212. doi: 10.5217/ir.2024.00135. Epub 2025 Feb 24. PMID 39988445